# A Phase 3, Open-label Study to Assess the Clinical Utility of Fluciclovine (18F) PET/CT in Patients with Prostate Cancer with Biochemical Recurrence after Radical Treatment

Blue Earth Diagnostics Study No: BED-004 Syne qua non Ltd Study No: BLS14004

# **Statistical Analysis Plan**

Version: Amendment 1 Final Date: 10<sup>th</sup> October 2018

#### For Syne qua non Ltd - Lead Statistician

-DocuSigned by:

Elizaleth Gardener



Signer Name: Elizabeth Gardener Signing Reason: I am the author of this document Signing Time: 10/11/2018 11:20:16 AM BST

-A40AC5551C6B49FBA379312B0D6DA509

#### For Blue Earth Diagnostics

DocuSigned by:

albert Chan



Signer Name: Albert Chau Signing Reason: I approve this document Signing Time: 10/11/2018 11:31:53 AM BST

-9E0EEC5DCDE944CCADBF63BA0CE6CA8E

Date: 10OCT2018 Version: Amendment 1 Final

# **Contents**

| 1 | INTRODUCTION | 5 |
|-------|--------------------------------------------|------|
| | GENERAL PRINCIPLES | |
| | STUDY OBJECTIVES AND DESIGN | |
| 3.1 | Study Objectives | |
| 3.2 | Study Design | |
| 3.3 | Visit Structure | |
| 3.4 | Sample Size | |
| 3.5 | Changes from the Protocol Planned Analysis | |
| | STUDY SUBJECTS | |
| 4.1 | Analysis sets | |
| 4.2 | Disposition of Subjects | |
| 4.3 | Protocol Deviations | |
| 4.4 | Background and Demographic Characteristics | |
| 4.4.1 | | |
| 4.4.2 | | |
| 4.4.3 | | |
| 4.4.4 | • | |
| 4.4.5 | | |
| 4.5 | Administration of Investigational Product | |
| 5 | EFFICACY EVALUATION | |
| 5.1 | Primary Efficacy Variable | |
| 5.2 | Secondary Efficacy Variables | 11 |
| 5.3 | Definition of Region Levels | |
| 5.4 | Statistical Analysis | |
| 5.4.1 | Primary Efficacy Analysis | 14 |
| 5.4.2 | Secondary Efficacy Analyses | . 18 |
| 5.4.3 | | |
| 5.4.4 | Interim Analyses and Data Monitoring | 19 |
| 5.4.5 | Examination of Subgroups | . 19 |
| 5.4.6 | Site Specific Sub-study | 19 |
| 6 | SAFETY EVALUATION | . 19 |
| 6.1 | Adverse Events | |
| 6.2 | Clinical Laboratory Evaluation | |
| 6.2.1 | Haematology | .21 |
| 6.2.2 | Biochemistry | .21 |
| 6.2.3 | - 1 | |
| 6.2.4 | - 17 | |
| 6.3 | Vital Signs | |
| 6.4 | Electrocardiography | |
| 7 | References | 22 |

# **ABBREVIATIONS**

| Abbreviation | Term |
|--------------|------------------------------------------------|
| AE | Adverse event |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| BCR | Biochemical recurrence |
| BMI | Body mass index |
| BUN | Blood urea nitrogen |
| CI | Confidence interval |
| CrCl | Creatinine clearance |
| CRF | Case report form |
| CT | Computerised Tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| EAS | Evaluable analysis set |
| ECG | Electrocardiogram |
| FAS | Full analysis set |
| GFR | Glomerular filtration rate |
| GGT | Gamma glutamyl transferase |
| LDH | Lactate dehydrogenase |
| MCH | Mean corpuscular hemoglobin |
| MCHC | Mean corpuscular hemoglobin concentration |
| MCV | Mean corpuscular volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | Magnetic resonance imaging |
| ms | Milliseconds |
| PCa | Prostate cancer |
| PET | Positron emission tomography |
| PPS | Per protocol set |
| PSA | Prostate specific antigen |
| PT | Preferred term |
| RBC | Red blood cell |
| RDW | Red cell distribution width |
| RP | Radical prostatectomy |
| RRT | Radical external beam radiotherapy |
| RT | Radiotherapy |
| SAE | Serious adverse event |
| SAF | Safety analysis set |
| SAP | Statistical analysis plan |
| SD | Standard deviation |

Syne qua non study no: BLS14004

Blue Earth Diagnostics study no: BED-004

SOC System organ class

TEAE Treatment emergent adverse event
TNM TNM classification of malignant tumours

WBC White blood cell

WHO World Health Organization

WHO DDE WHO Drug Dictionary Enhanced


#### 1 INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the final protocol version dated 24<sup>th</sup> March 2015 and amendments 1-4 dated 30<sup>th</sup> November 2015, 5<sup>th</sup> April 2016, 2<sup>nd</sup> March 2017 and 4<sup>th</sup> June 2018.

The SAP describes the tables, listings and figures which will be provided upon completion of the study. The SAP will be finalised before locking the database.

The table, listing and figure shells will be supplied in a separate document.

#### 2 GENERAL PRINCIPLES

The analysis and statistical reporting will be conducted at Syne qua non using SAS version 9.2 or higher.

All listings will be based on all enrolled subjects unless specified otherwise. All tables will be presented by site and overall for the appropriate analysis population.

Descriptive summary statistics for continuous variables will include number of subjects (n), mean, standard deviation (SD), minimum, median, and maximum, unless specified otherwise. The precision of these summary statistics is defined in the table, figure and listing shells document.

Descriptive summary statistics for categorical variables will include frequency counts and percentages [n (%)]. Unless stated otherwise, the denominator for percentage calculations will be the number of subjects in the analysis set.

For treatment response baseline prostate specific antigen (PSA) is the most recent PSA measurement prior to salvage therapy for subjects who had salvage treatment and the most recent PSA measurement prior to the 18F-fluciclovine positron emission tomography/computerised tomography (PET/CT) for non-salvage subjects. If no PSA measurement is available just prior to salvage therapy, baseline will be defined as the most recent PSA measurement prior to fluciclovine (<sup>18</sup>F) scan. For all other variables, and for baseline PSA other than for treatment response, baseline is defined as the most recent value prior to fluciclovine (<sup>18</sup>F) administration.

In general, there will be no imputation of missing data, however where dates are partially missing dates may be imputed for calculation purposes, details are given under relevant section.

#### 3 STUDY OBJECTIVES AND DESIGN

# 3.1 Study Objectives

The primary objective of the study is to confirm the clinical benefit of fluciclovine (<sup>18</sup>F) PET/CT in affecting management decisions in subjects with biochemical recurrence (BCR) being considered for radical salvage treatment (with curative intent).

The secondary objectives of the study are

 To assess possible improvement in outcome of radical salvage treatment based on fluciclovine (<sup>18</sup>F) PET/CT being included in the assessment


- To assess the PSA threshold for positive lesion detection by fluciclovine (<sup>18</sup>F) PET/CT in BCR
- To assess the safety of fluciclovine (<sup>18</sup>F) injection in subjects undergoing PET/CT

# 3.2 Study Design

This will be an open-labelled, multi-centred study in the United Kingdom.

The study group will include up to 180 subjects with a diagnosis of BCR of previous radically treated prostate cancer (PCa), and who are being considered for radical salvage therapy.

Subjects will have a fluciclovine (<sup>18</sup>F) PET/CT scan in addition to standard work-up for radical salvage therapy. The clinical utility of fluciclovine (<sup>18</sup>F) PET/CT will be assessed by recording changes to the recommended management plan influenced by the scan result.

The summary flow chart of the study design is as follows:



#### 3.3 Visit Structure

The visit structure and scheduled assessments are detailed in Appendix A: Schedule of study procedures of the protocol.


### 3.4 Sample Size

For the primary objective of treatment change evaluation, a minimum of 171 subjects with complete primary endpoint data will be required to allow for a width of +/-6% in a two-sided 95% confidence interval (CI). This is based on the conservative assumption that 20% of subjects will have a treatment change, as fluciclovine (<sup>18</sup>F) PET/CT has been shown to upstage 25.7% of subjects with recurrent prostate cancer, and also based on the management change studies reported on choline PET/CT. The aim is to recruit 180 subjects for this trial, based on an anticipated primary endpoint drop-out rate of 5%.

### 3.5 Changes from the Protocol Planned Analysis

The protocol specified "Improvement in outcome of radical salvage treatment based on fluciclovine (18F) PET/CT being included in the assessment" as a secondary endpoint. This was to be assessed based on PSA and radiological response. Due to lack of data being recorded for radiological response this definition was not used, treatment response was instead assessed using PSA only (see section 5.4.2.1.).

#### 4 STUDY SUBJECTS

### 4.1 Analysis sets

The list of subjects to be included in each of the analysis set is to be agreed between the Syne qua non statistician and Blue Earth Diagnostics once all study data are available and prior to database lock.

Enrolled Set: All subjects who entered screening.

**Safety Analysis Set (SAF)**: All subjects who have been included in the database and have been administered fluciclovine (<sup>18</sup>F) will be included in the Safety Analysis Set (SAF).

**Full Analysis Set (FAS)**: All subjects enrolled who have had a fluciclovine (<sup>18</sup>F) PET/CT scan will be included in the Full Analysis Set (FAS).

**Evaluable Analysis Set (EAS)**: All subjects from the FAS who have an intended treatment management plan completed and a revised management plan page completed will be included in the Evaluable Analysis Set (EAS).

**Per Protocol Set (PPS)**: All subjects in the EAS without major significant deviation following review of the protocol deviation list.

# 4.2 Disposition of Subjects

The number and percentage of all subjects enrolled, included in each analysis set, who completed the study and who prematurely withdrew, including a breakdown of the primary reasons for withdrawal, will be presented.

All enrolled subjects will be listed indicating their membership to the evaluable analysis set along with the reason for exclusion.

Completion and withdrawal information will be listed, including individual reasons for withdrawal.


#### 4.3 Protocol Deviations

Failed inclusion criteria and failed exclusion criteria will be listed for screening failures.

The number and percentage of subjects within each deviation category will be presented by deviation type (Major Significant, Major or Minor) and by site and overall. The deviation category and type will be provided by Blue Earth Diagnostics. All protocol deviations will be listed.

## 4.4 Background and Demographic Characteristics

#### 4.4.1 Demographic and Baseline Characteristics

Demographic characteristics (age, ethnic origin and race collected at Screening), body measurements (height, weight collected, and BMI derived at Visit 2) will be summarised for the enrolled set, FAS, EAS and PPS populations.

Body mass index (BMI) is calculated as (weight (kg)/height (m)<sup>2</sup>).

Individual demographic characteristics and body measurements data will be listed.

#### 4.4.2 Medical History

Medical history events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 18.1.

The number and percentage of subjects from the FAS with previous medical history and current events will be tabulated by system organ class (SOC), preferred term (PT). SOCs will be ordered in decreasing frequency of the total number of subjects with medical history events reported in each SOC and PTs will be ordered within a SOC in decreasing frequency of the total number of subjects with each medical history event. This table will be repeated for all events, regardless of whether previous or current events.

All medical history events will be listed.

#### 4.4.3 Prostate Cancer History

Details of prostate cancer history will be summarised for subjects from the FAS, and will consist of:

- Time since initial diagnosis (months), calculated as [12\*(date of informed consent date of initial prostate cancer diagnosis + 1)/365.25]
- TNM stage: Pathological TNM stage if available, otherwise Clinical TNM stage. A summary for T1 total, T2 total and T3 total will be provided as the sum of the number of subjects in each of the subgroups plus any subjects where only T1, T2 or T3 was recorded.
- Gleason total score: Gleason total score from surgery if available, otherwise Gleason total score from biopsy
- Time since adjuvant treatment (months), calculated as [12\*(date of informed consent stop date of adjuvant treatment + 1)/365.25]
- Duration of adjuvant treatment (months), calculated as [12\*(stop date of adjuvant treatment – start date of adjuvant treatment + 1)/365.25]

- Time since diagnosis of biochemical recurrence (days), calculated as (date of informed consent – date of diagnosis of biochemical recurrence + 1). Time since diagnosis of BCR may be derived in months if more appropriate.
- Baseline PSA value
- Baseline PSA category (0 0.2, >0.2 0.5, >0.5 1, >1 2, >2 5, >5 10 and >10)

In addition, summary table to summarise baseline Prostate Specific Antigen (PSA) by Prior Radical Prostatectomy status (Prior Radical Prostatectomy vs No Prior Radical Prostatectomy) using descriptive statistics (number of subjects (n), mean, standard deviation (SD), minimum, median, and maximum), will be produced.

Details of prostate cancer history will be listed.

Date imputation for incomplete dates:

- If day part missing, put 15<sup>th</sup> of the month
- If day and month parts missing, put 01 July

#### 4.4.4 Cancer Therapies for Prostate Cancer

Cancer therapies for prostate cancer will be coded according to the World Health Organization Drug Dictionary Enhanced (WHO DDE) (Enhanced) version Sep 2015.

Cancer therapies will be categorised as follows:

Subjects with radical prostatectomy:

- Radiotherapy
- No radiotherapy

Subjects without radical prostatectomy:

- Radiotherapy only
  - o EBRT only
  - Brachytherapy only
  - EBRT and brachytherapy
- Radiotherapy and other therapies
  - EBRT and other therapies
  - Brachytherapy and other therapies
- Other therapies

Prior cancer therapies for prostate cancer are defined as those for which the end date is prior to the date of injection of fluciclovine (<sup>18</sup>F).

Concomitant/post-scan cancer therapies for prostate cancer are defined as those with a start date on or after the injection date of fluciclovine (<sup>18</sup>F), or those with a start date before the injection date of fluciclovine (<sup>18</sup>F) but which continued with a stop on or after the injection date of fluciclovine (<sup>18</sup>F). Summaries for subjects with prior and post-scan radical prostatectomy will be presented separately.


Summary table to summarise time from <sup>18</sup>F-fluciclovine PET/CT to first post-<sup>18</sup>F-fluciclovine treatment in days using descriptive statistics (number of subjects (n), mean, SD, minimum, median, and maximum) will be provided.

If cancer therapy dates are incomplete and it is not clear whether the medication was concomitant, it will be assumed to be concomitant.

The number and percentage of subjects per category of prostate cancer therapy will be presented for all subjects from the SAF, separately for subjects with and without radical prostatectomy. This summary will be repeated for prior and concomitant cancer therapies.

All therapies for prostate cancer will be listed including type of therapy, reported therapy name, medication class, standardised medication name, dose, dose unit, route of administration, start date and end date or 'ongoing' flag, therapy comments.

#### 4.4.5 Prior and Concomitant Medications

Prior and concomitant medications will be coded according to the World Health Organization Drug Dictionary Enhanced (WHO DDE) (Enhanced) version Sep 2015.

Prior medications are defined as those for which the end date is prior to the date of injection of fluciclovine (18F).

Concomitant medications are defined as those with a start date on or after the injection date of fluciclovine (<sup>18</sup>F), or those with a start date before the injection date of fluciclovine (<sup>18</sup>F) but which continued with a stop date on or after the injection date of fluciclovine (<sup>18</sup>F).

If medication dates are incomplete and it is not clear whether the medication was concomitant, it will be assumed to be concomitant.

The number and percentage of subjects who took any medications will be presented by centre and overall by medication class, standardised medication names sorted alphabetically for all subjects from the SAF, separately for prior medications and concomitant medications.

All prior and concomitant medications will be listed including reported name, medication class, standardised medication name, indication, dose, dose unit, frequency, route of administration, start date and end date or 'ongoing' flag.

# 4.5 Administration of Investigational Product

The volume of undiluted fluciclovine, activity of fluciclovine and injection site reaction during and following fluciclovine administration will be summarised for subjects in the SAF.

#### 5 EFFICACY EVALUATION

All listings will be based on the FAS unless specified otherwise. The primary efficacy analysis will be based on the EAS and will be repeated on the PPS as a secondary analysis. The secondary efficacy analyses will be based on the FAS.


#### 5.1 **Primary Efficacy Variable**

The primary efficacy variable is the record of the revised management plan post fluciclovine (<sup>18</sup>F) PET/CT scan in comparison to the pre-scan intended management plan.

#### 5.2 **Secondary Efficacy Variables**

The secondary efficacy variables are:

- The proportion of subjects who have a sustained response to radical salvage therapy.
- PSA levels in relation to scan positivity will be analysed to determine the optimal PSA threshold for detecting recurrent PCa by fluciclovine (18F) PET/CT.

# **Definition of Region Levels**

Two main regions will be analysed, the prostate and prostate bed and the extraprostatic region.

The prostate and prostate bed include the following lesion locations:

- Prostate bed left
- Prostate bed right
- Peripheral zone left
- Peripheral zone right
- Central gland left
- Central gland right
- Left seminal vesicle
- Right seminal vesicle

The extra-prostatic regions include the following lesion locations

- Lymph nodes
  - Pelvic lymph nodes
    - Common iliac left
    - Common iliac right
    - Internal iliac left
    - Internal iliac right
    - External iliac left
    - External iliac right
    - Obturator left
    - Obturator right
    - Pre-sacral left

- Pre-sacral right
- Peri-rectal anterior
- Peri-rectal posterior
- Peri-rectal left
- Peri-rectal right
- Inguinal left
- Inguinal right

- Retroperitoneal lymph nodes
  - Para-aortic
  - Retro-aortic
  - Para-caval
  - Retro-caval
- Other lymph nodes
  - Intra-peritoneal
  - Mediastinal left
  - Mediastinal right
  - Axillary left
- Soft tissues/parenchyma
  - o Lung upper lobe left
  - Lung upper lobe right
  - Lung middle lobe right
  - Lung lower lobe left
  - o Lung lower lobe right
  - Brain left
  - o Brain right
  - Liver left
  - Liver right
  - Spleen
  - Subcutaneous/cutaneous
  - Muscle
  - Bowel
- Bones
  - o Skull
    - Skull base/maxilla left
    - Skull base/maxilla right
    - Mandible left
    - Mandible right
  - Vertebra
    - Vertebra C1
    - Vertebra C2
    - Vertebra C3
    - Vertebra C4

- Aorto-caval
- Retrocrural left
- Retrocrural right
- Axillary right
- Cervical left
- Cervical right

Vertebra C5

Vertebra C6

Vertebra C7

Vertebra T1

- Vertebra T2
- Vertebra T3
- Vertebra T4
- Vertebra T5
- Vertebra T6
- Vertebra T7
- Vertebra T8
- Vertebra T9
- Vertebra T10
- Vertebra T11

#### o Chest

- 1<sup>st</sup> rib left
- 1st rib right
- 2<sup>nd</sup> rib left
- 2<sup>nd</sup> rib right
- 3<sup>rd</sup> rib left
- 3<sup>rd</sup> rib right
- 4<sup>th</sup> rib left
- 4<sup>th</sup> rib right
- 5<sup>th</sup> rib left
- 5<sup>th</sup> rib right
- 6<sup>th</sup> rib left
- 6<sup>th</sup> rib right
- 7<sup>th</sup> rib left
- 7<sup>th</sup> rib right
- 8<sup>th</sup> rib left

#### Pelvis

- Ilium left
- Ilium right
- Superior pubic ramus left
- Superior pubic ramus right
- Inferior pubic ramus left

- Vertebra T12
- Vertebra L1
- Vertebra L2
- Vertebra L3
- Vertebra L4
- Vertebra L5
- Sacrum left
- Sacrum right
- Sacrum central
- 8<sup>th</sup> rib right
- 9<sup>th</sup> rib left
- 9<sup>th</sup> rib right
- 10<sup>th</sup> rib left
- 10<sup>th</sup> rib right
- 11<sup>th</sup> rib left
- 11<sup>th</sup> rib right
- 12<sup>th</sup> rib left
- 12<sup>th</sup> rib right
- Sternum
- Clavicle left
- Clavicle right
- Scapula left
- Scapula right
- Inferior pubic ramus right
- Pubic body left
- Pubic body right
- Ischium left
- Ischium right

#### Appendicular

- Proximal humerus left
- Proximal humerus right
- Proximal femur left
- Proximal femur right

# 5.4 Statistical Analysis

#### **5.4.1 Primary Efficacy Analysis**

The analysis of the primary outcome will be performed on the EAS as the primary analysis and will be repeated on the PPS as a secondary analysis. Comparisons between the original treatment plan and the revised treatment plan will be categorised as no change, major change or other change. The definitions of the change categories are listed below.

- No change: the original treatment plan is the same as the revised treatment plan
- Major change: the original treatment plan is not the same as the revised treatment plan and the grouping for the original treatment plan is not the same as the grouping for the revised treatment plan

These will be further split and presented according to the following categories:

- Salvage or Non-curative systemic therapy to Watchful waiting
- Salvage therapy to Non-curative systemic therapy
- Non-curative systemic therapy to Salvage therapy
- Alternative Major change
- Other change: the original treatment plan is not the same as the revised treatment plan but the grouping for the original treatment plan is the same as the grouping for the revised treatment plan

These will be further split and presented according to the following categories:

- Modified RT field plan
- Modified androgen-deprivation regimen
- Alternative Other change

Groupings of treatment plans are detailed in the following table:


Version: Amendment 1 Fina ST/form/010/6

| Original Treatment<br>Plan | Grouping for<br>Original Tx Plan | Revised Treatment | Grouping for<br>Revised Tx Plan |
|---|---|---|---|
| Was androgen deprivation therapy planned | Androgen<br>Deprivation<br>Therapy | Androgen deprivation therapy | Androgen<br>deprivation therapy |
| | | Watch and wait | Watch and wait |
| | | Chemotherapy | Chemotherapy |
| Salvage<br>radiotherapy to the<br>prostate bed | | Salvage radiotherapy to the prostate bed | |
| Salvage radiotherapy to the prostate bed, with boost to areas guided by conventional imaging | Salvage<br>Radiotherapy | Salvage radiotherapy to the prostate bed, with boost to areas guided by conventional imaging | Salvage<br>Radiotherapy |
| | | Salvage radiotherapy to the prostate bed with boost to areas guided by fluciclovine (18F) PET/CT | |
| Salvage<br>radiotherapy to the<br>prostate bed and<br>whole pelvis | | Salvage<br>radiotherapy to the<br>prostate bed and<br>whole pelvis | |
| Salvage radiotherapy to the prostate bed and whole pelvis, with boost to areas guided by conventional imaging | Salvage<br>Radiotherapy | Salvage radiotherapy to the prostate bed and whole pelvis, with boost to areas guided by conventional imaging | Salvage<br>Radiotherapy |
| | | Salvage radiotherapy to the prostate bed and whole pelvis with boost to areas guided by fluciclovine (18F) PET/CT | |

| Original Treatment<br>Plan | Grouping for<br>Original Tx Plan | Revised Treatment Plan | Grouping for<br>Revised Tx Plan |
|---|---|---|---|
| Salvage<br>cryotherapy | | Salvage<br>cryotherapy | |
| | Salvage<br>Cryotherapy | Salvage cryotherapy with boost to areas guided by fluciclovine (18F) PET/CT | Salvage<br>Cryotherapy |
| Salvage<br>brachytherapy | | Salvage<br>brachytherapy | |
| | Salvage<br>Brachytherapy | Salvage brachytherapy with boost to areas guided by fluciclovine (18F) PET/CT | Salvage<br>Brachytherapy |
| | | Salvage brachytherapy with treatment plan guided by fluciclovine (18F) PET/CT | |
| Salvage HIFU | | Salvage HIFU | |
| | Salvage HIFU | Salvage HIFU with treatment plan guided by fluciclovine (18F) PET/CT | Salvage HIFU |
| Salvage prostatectomy | | Salvage prostatectomy | |
| | Salvage<br>Prostatectomy | Salvage prostatectomy with targeted resection / sampling of fluciclovine (18F) positive areas outside conventional surgical field | Salvage<br>Prostatectomy |
| Salvage<br>prostatectomy and<br>limited lymph node<br>dissection | | Salvage<br>prostatectomy and<br>limited lymph node<br>dissection | |

| Original Treatment<br>Plan | Grouping for<br>Original Tx Plan | Revised Treatment<br>Plan | Grouping for<br>Revised Tx Plan |
|---|---|---|---|
| | | Salvage prostatectomy and limited lymph node dissection with targeted resection / sampling of fluciclovine (18F) positive areas outside surgical field | |
| Salvage prostatectomy and extended lymph node dissection (including internal and external iliac, and obturator nodes) | | Salvage prostatectomy and extended lymph node dissection (including internal and external iliac, and obturator nodes) | |
| | | Salvage prostatectomy and extended lymph node dissection (including internal and external iliac, and obturator nodes) with targeted resection / sampling of fluciclovine (18F) positive areas outside surgical field | |
| | | Targeted salvage treatment of fluciclovine (18F) positive extra-pelvic / bony areas | Targeted salvage<br>treatment |
| | | Other | Other |

The classification and sub-classification of change in treatment management plan will be agreed prior to data base lock.

The number, percentage and exact 95% CI of subjects with and without a change in management plan after the fluciclovine (18F) scan results become available will be presented. In addition, the number and percentage of subjects with changes categorised as major or other will be presented. These summaries will be repeated separately for subjects with a positive and a negative fluciclovine (18F) scan and for subjects without prostatectomy and with prostatectomy.

The number, percentage and 95% CI of subjects who agreed to the revised management plan after fluciclovine (<sup>18</sup>F) scan results become available will be presented.

Details of the intended management plan, revised management plan and agreed management plan will be listed.

#### 5.4.2 Secondary Efficacy Analyses

#### 5.4.2.1 Treatment response as assessed by change in PSA

An assessment of treatment response, which is based on the percentage change in PSA from baseline to the last value reported, is defined as:

- >=30% decrease in PSA will be considered to be a response to treatment
- <25% increase or <30% decrease will be classified as stable disease</li>
- >=25% increase in PSA will be classified as disease progression

See section 2 General Principles for baseline definition.

The number, percentage and exact 95% CI of subjects having a treatment response, stable disease and disease progression, as assessed by change in PSA, will be presented overall and separately for subjects in the FAS who had salvage treatment, for subjects who had non-salvage treatment, for those with a change in management plan and for subjects with no change in management plan following the <sup>18</sup>F-fluciclovine PET/CT scan. In addition, treatment response assessed by change in PSA will be summarised by disease location (local disease versus extra-prostatic disease) and treatment administered.

The percentage change in PSA from baseline to the last value reported will be summarised overall and by subjects who had a change in management plan versus those who did not have a change in management plan following the <sup>18</sup>F-fluciclovine PET/CT scan, disease location and treatment administered.

Finally, a waterfall plot of the maximum percentage reduction in PSA during the 4-8 month window will be presented on the y-axis and each subject will be represented by a bar on the x-axis. The bars will be ordered in descending order of the magnitude of the percentage change in PSA value.

Treatment response and the factors used to assess the response will be listed in full.

#### 5.4.2.2 PSA threshold

The detection rate (DR) will be calculated as number of positive fluciclovine (<sup>18</sup>F) scan results/total number of scans.


The point estimate (expressed in percentage) of the DR will be presented at the region level and at the subject level. These rates will be presented for all subjects from the FAS and PPS, overall and across a range of baseline PSA values:

- 0 0.2
- $\bullet$  >0.2 0.5
- $\bullet$  >0.5 1.0
- $\bullet$  >1.0 2.0
- $\bullet$  >2.0 5.0
- $\bullet$  >5.0 10.0
- >10.0

to determine the optimum PSA threshold for lesion detection. See section 2 General Principles for baseline definition.

The detection rates will also be summarised across the following baseline Gleason score categories: <=6, 7, 8 and >=9.

All fluciclovine (18F) and other imaging results will be listed.

#### **Handling of Dropouts or Missing Data** 5.4.3

Subjects who withdrew from the study prior to completion will be summarised. Withdrawn subjects will not be directly replaced and no imputation of missing data will be conducted.

#### 5.4.4 **Interim Analyses and Data Monitoring**

A single interim analysis of the primary endpoint will be performed in the first 85 evaluable subjects. If the number of treatment changes is greater than 45 (52.9%, with a 97.5% two-sided CI of 40.3%-62.3%, so the lower limit is over 40%), the trial will be terminated early due to overwhelming effectiveness. If the number of treatment changes is 8 or fewer (9.4%, with a 97.5% two-sided CI of 3.6%-18.9%, so the upper limit in this population is below the 20% of the null hypothesis), the trial will be terminated early due to futility.

#### **Examination of Subgroups**

No subgroup analyses will be conducted during the study.

#### **Site Specific Sub-study** 5.4.6

A site specific sub-study will be conducted in order to compare the ordered subset expectation maximisation (OSEM) standard of care method of reconstructing PET/CT images with that of the Bayesian penalised likelihood method of PET/CT image reconstruction. The analysis of the sub-study results is beyond the scope of this SAP.

#### SAFETY EVALUATION

All safety evaluations will be performed on the safety analysis set (SAF) unless specified otherwise.


All safety tables will be presented by centre and overall.

Subjects will be included and counted in summary tables only if they have available data.

#### 6.1 Adverse Events

Adverse events (AE) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 17.1.

A treatment-emergent adverse event (TEAE) is defined as an AE with start date/time on or after the start/time of fluciclovine (<sup>18</sup>F) administration, or AEs with worsening intensity on or after the start date/time of fluciclovine (<sup>18</sup>F) administration.

AEs with unknown start date/time will be assumed to be treatment-emergent unless the end date/time is known to be before the fluciclovine (<sup>18</sup>F) administration.

Summary tables will be produced for all TEAEs occurring up to 42 days (i.e. occurring between day 1 and day 43) after the fluciclovine (<sup>18</sup>F) administration.

An overall summary of TEAEs will be created including:

- number of TEAEs and number of subjects with TEAEs,
- number of TEAEs and number of subjects with TEAEs associated with the injection site,
- number of serious TEAEs and number of subjects with serious TEAEs,
- number of subjects with TEAEs by CTCAE grade (Grade 1 to Grade 5),
- number of subjects with TEAEs by relationship to fluciclovine (unrelated, possibly related, probably related, definitely related and related, where related adverse events are those classified as possibly, probably and definitely related to fluciclovine <sup>18</sup>F)

The number and percentage of subjects experiencing TEAEs will be presented by system organ class (SOC) and preferred term (PT). System organ class and preferred term will be presented in decreasing frequency of the total number of subjects with TEAEs. If a subject experienced more than one treatment-emergent adverse event, the subject will be counted once for each system organ class and once for each preferred term.

The number and percentage of subjects experiencing TEAEs will be presented by SOC, PT and CTCAE grade. SOC and PT will be presented in decreasing frequency of the total number of subjects with TEAEs. If a subject experienced more than one TEAE, the subject will be counted once for each SOC and once for each PT at the worst severity.

The number and percentage of subjects experiencing TEAEs will be presented by SOC, PT and relationship to study drug. SOC and PT will be presented in decreasing frequency of the total number of subjects with TEAEs. If a subject experienced more than one TEAE, the subject will be counted once for each SOC and once for each PT at the closest relationship to study drug.

All adverse events will be listed and TEAEs will be identified. AEs occurring up to 42 days after fluciclovine (<sup>18</sup>F) administration will be flagged. All SAEs will be listed separately.


### 6.2 Clinical Laboratory Evaluation

#### 6.2.1 Haematology

Haematology values will be summarised by parameter and visit, and also for change from baseline (last pre-scan value vs first post-scan value).

All haematology values will be listed showing reference ranges (flagging abnormal findings).

#### 6.2.2 Biochemistry

Biochemistry values will be summarised by parameter and visit, and also for change from baseline (last pre-scan value vs first post-scan value).

Additionally, from the serum creatinine levels (mg/dL), creatinine clearance (CrCl) will be derived using the Cockcroft Gault formula (Cockroft DW, 1976) and the glomerular filtration rate (GFR) will be derived using the MDRD formula (Levey AS, 2006) as follows:

- Cockcroft-Gault formula: CrCl (mL/min) = [(140 age) \* (Weight in kg) \* (0.85 if female)] / (72 \* Creatinine)
- MDRD formula: GFR (mL/min) = 175 \* Creatinine<sup>-1.154</sup> \* age<sup>-0.203</sup> \* (1.212 if subject is black) \* (0.742 if female)

CrCl and GFR categories (≤30 mL/min, >30 - ≤60, >60 - ≤90, >90 mL/min) will be summarised by time window, and the shift table of baseline status against the worst status on or after fluciclovine (¹8F) administration will be presented.

All biochemistry values will be listed showing reference ranges and flagging abnormal findings.

#### 6.2.3 Urinalysis dipstick

All urinalysis results will be listed.

#### 6.2.4 Urine microscopy

All urine microscopy results will be listed.

# 6.3 Vital Signs

Vital signs include pulse rate, systolic and diastolic blood pressure.

Vital sign values will be summarised by parameter and time point, and also for change from baseline.

Details of vital signs data will be listed.

# 6.4 Electrocardiography

Electrocardiogram (ECG) interpretation is recorded at screening and visit 4.

ECG interpretations will be summarised by shift tables highlighting any changes between screening and visit 4.


#### 7 REFERENCES

- Cockroft DW, G. M. (1976). Prediction of creatinine clearance from serum creatinine. *Nephron*, 31-41.
- Levey AS, C. J. (2006). Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. *Ann Intern Med*, 247-254.




**Certificate Of Completion** 

Envelope Id: 93B644B8A8914520914F18451BC4D479

Subject: BED004 (BLS14004): Statistical Analysis Plan Amendment 1 for signature

Source Envelope:

Document Pages: 22Signatures: 2Envelope Originator:Certificate Pages: 5Initials: 0Elizabeth GardenerAutoNav: EnabledGostling HouseEnvelopeld Stamping: EnabledDiss Business Park

Time Zone: (UTC) Dublin, Edinburgh, Lisbon, London Diss, Norfolk IP22 4GT

elizabeth.gardener@synequanon.com

IP Address: 62.232.1.93

Sent: 10/11/2018 11:19:15 AM

Viewed: 10/11/2018 11:19:49 AM

Signed: 10/11/2018 11:20:20 AM

Sent: 10/11/2018 11:20:21 AM

Viewed: 10/11/2018 11:31:22 AM

Signed: 10/11/2018 11:31:58 AM

Status: Completed

**Record Tracking** 

Status: Original Holder: Elizabeth Gardener Location: DocuSign

10/11/2018 11:13:39 AM elizabeth.gardener@synequanon.com

Signer Events Signature Timestamp

Elizabeth Gardener

Elizabeth Gardener

elizabeth.gardener@synequanon.com

Senior Statistician Syne qua non

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

A40AC555-1C6B-49FB-A379-312B0D6DA509

Using IP Address: 62.232.1.93

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I am the author of this document

**Electronic Record and Signature Disclosure:** 

Not Offered via DocuSign

Albert Chau

albert@datacision.co.uk

Director

**Datacision Limited** 

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

albert Chan

9E0EEC5D-CDE9-44CC-ADBF-63BA0CE6CA8E

Using IP Address: 92.40.249.236

Signed using mobile

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 10/11/2018 11:31:22 AM

ID: 7c339459-f310-4678-b276-cd05df73f47d

In Person Signer Events Signature Timestamp

Editor Delivery Events Status Timestamp

Agent Delivery Events Status Timestamp

Intermediary Delivery Events Status Timestamp

| Certified Delivery Events | Status | Timestamp |
|---|---|---|
| Carbon Copy Events | Status | Timestamp |
| Corinne Hedgley Corinne.Hedgley@synequanon.com Senior Project Manager Syne qua non Ltd | COPIED | Sent: 10/11/2018 11:31:59 AM |

Security Level: Email, Account Authentication (Required)

**Electronic Record and Signature Disclosure:**Not Offered via DocuSign

| Notary Events | Signature | Timestamp |
|---|---|---|
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 10/11/2018 11:31:59 AM |
| Certified Delivered | Security Checked | 10/11/2018 11:31:59 AM |
| Signing Complete | Security Checked | 10/11/2018 11:31:59 AM |
| Completed | Security Checked | 10/11/2018 11:31:59 AM |
| Payment Events Status Timestamps | | |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Syne qua non Ltd (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through your DocuSign, Inc. (DocuSign) Express user account. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to these terms and conditions, please confirm your agreement by clicking the 'I agree' button at the bottom of this document.

#### **Getting paper copies**

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. For such copies, as long as you are an authorized user of the DocuSign system you will have the ability to download and print any documents we send to you through your DocuSign user account for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

## Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

#### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. To indicate to us that you are changing your mind, you must withdraw your consent using the DocuSign 'Withdraw Consent' form on the signing page of your DocuSign account. This will indicate to us that you have withdrawn your consent to receive required notices and disclosures electronically from us and you will no longer be able to use your DocuSign Express user account to receive required notices and consents electronically from us or to sign electronically documents from us.

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through your DocuSign user account all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### **How to contact Syne qua non Ltd:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: pauline.allen@synequanon.com

#### To advise Syne qua non Ltd of your new e-mail address

To let us know of a change in your e-mail address where we should send notices and disclosures electronically to you, you must send an email message to us at Pauline.Allen@synequanon.com and in the body of such request you must state: your previous e-mail address, your new e-mail address. We do not require any other information from you to change your email address.. In addition, you must notify DocuSign, Inc to arrange for your new email address to be reflected in your DocuSign account by following the process for changing e-mail in DocuSign.

### To request paper copies from Syne qua non Ltd

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an e-mail to Pauline.Allen@synequanon.com and in the body of such request you must state your e-mail address, full name, US Postal address, and telephone number. We will bill you for any fees at that time, if any.

### To withdraw your consent with Syne qua non Ltd

To inform us that you no longer want to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your DocuSign account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may; ii. send us an e-mail to pauline.allen@synequanon.com and in the body of such request you must state your e-mail, full name, IS Postal Address, telephone number, and account number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

| Operating Systems: | Windows2000? or WindowsXP? |
|----------------------------|----------------------------------------------|
| Browsers (for SENDERS): | Internet Explorer 6.0? or above |
| Browsers (for SIGNERS): | Internet Explorer 6.0?, Mozilla FireFox 1.0, |
| | NetScape 7.2 (or above) |
| Email: | Access to a valid email account |
| Screen Resolution: | 800 x 600 minimum |
| Enabled Security Settings: | •Allow per session cookies |
| | •Users accessing the internet behind a Proxy |
| | Server must enable HTTP 1.1 settings via |
| | proxy connection |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an email message at the email address we have on file for you at that time providing you with the revised hardware and software requirements, at which time you will have the right to withdraw your consent.

#### Acknowledging your access and consent to receive materials electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please verify that you were able to read this electronic disclosure and that you also were able to print on paper or electronically save this page for your future reference and access or that you were able to e-mail this disclosure and consent to an address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format on the terms and conditions described above, please let us know by clicking the 'I agree' button below.

By checking the 'I Agree' box, I confirm that:

- I can access and read this Electronic CONSENT TO ELECTRONIC RECEIPT OF ELECTRONIC RECORD AND SIGNATURE DISCLOSURES document; and
- I can print on paper the disclosure or save or send the disclosure to a place where I can print it, for future reference and access; and
- Until or unless I notify Syne qua non Ltd as described above, I consent to receive from exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to me by Syne qua non Ltd during the course of my relationship with you.

# A Phase 3, Open-label Study to Assess the Clinical Utility of Fluciclovine (18F) PET/CT in Patients with Prostate Cancer with Biochemical Recurrence after Radical Treatment

Blue Earth Diagnostics Study No: BED-004 Syne qua non Ltd Study No: BLS14004

# **Statistical Analysis Plan**

Version: Amendment 1 Final Date: 10<sup>th</sup> October 2018

#### For Syne qua non Ltd - Lead Statistician

-DocuSigned by:

Elizabeth Gardener



Signer Name: Elizabeth Gardener Signing Reason: I am the author of this document Signing Time: 10/11/2018 11:20:16 AM BST

-A40AC5551C6B49FBA379312B0D6DA509

#### For Blue Earth Diagnostics

DocuSigned by:

Albert Chan



Signer Name: Albert Chau Signing Reason: I approve this document Signing Time: 10/11/2018 11:31:53 AM BST

-9E0EEC5DCDE944CCADBF63BA0CE6CA8E


# **Contents**

| 1 | INTRODUCTION | 5 |
|-------|--------------------------------------------|------|
| | GENERAL PRINCIPLES | |
| | STUDY OBJECTIVES AND DESIGN | |
| 3.1 | Study Objectives | |
| 3.2 | Study Design | |
| 3.3 | Visit Structure | |
| 3.4 | Sample Size | |
| 3.5 | Changes from the Protocol Planned Analysis | |
| | STUDY SUBJECTS | |
| 4.1 | Analysis sets | |
| 4.2 | Disposition of Subjects | |
| 4.3 | Protocol Deviations | |
| 4.4 | Background and Demographic Characteristics | |
| 4.4.1 | | |
| 4.4.2 | | |
| 4.4.3 | | |
| 4.4.4 | • | |
| 4.4.5 | | |
| 4.5 | Administration of Investigational Product | |
| 5 | EFFICACY EVALUATION | |
| 5.1 | Primary Efficacy Variable | |
| 5.2 | Secondary Efficacy Variables | 11 |
| 5.3 | Definition of Region Levels | |
| 5.4 | Statistical Analysis | |
| 5.4.1 | Primary Efficacy Analysis | 14 |
| 5.4.2 | Secondary Efficacy Analyses | . 18 |
| 5.4.3 | | |
| 5.4.4 | Interim Analyses and Data Monitoring | 19 |
| 5.4.5 | Examination of Subgroups | . 19 |
| 5.4.6 | Site Specific Sub-study | 19 |
| 6 | SAFETY EVALUATION | . 19 |
| 6.1 | Adverse Events | |
| 6.2 | Clinical Laboratory Evaluation | |
| 6.2.1 | Haematology | .21 |
| 6.2.2 | Biochemistry | .21 |
| 6.2.3 | - 1 | |
| 6.2.4 | - 17 | |
| 6.3 | Vital Signs | |
| 6.4 | Electrocardiography | |
| 7 | References | 22 |

# **ABBREVIATIONS**

| Abbreviation | Term |
|--------------|------------------------------------------------|
| AE | Adverse event |
| ALT | Alanine aminotransferase |
| AST | Aspartate aminotransferase |
| BCR | Biochemical recurrence |
| BMI | Body mass index |
| BUN | Blood urea nitrogen |
| CI | Confidence interval |
| CrCl | Creatinine clearance |
| CRF | Case report form |
| CT | Computerised Tomography |
| CTCAE | Common Terminology Criteria for Adverse Events |
| EAS | Evaluable analysis set |
| ECG | Electrocardiogram |
| FAS | Full analysis set |
| GFR | Glomerular filtration rate |
| GGT | Gamma glutamyl transferase |
| LDH | Lactate dehydrogenase |
| MCH | Mean corpuscular hemoglobin |
| MCHC | Mean corpuscular hemoglobin concentration |
| MCV | Mean corpuscular volume |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | Magnetic resonance imaging |
| ms | Milliseconds |
| PCa | Prostate cancer |
| PET | Positron emission tomography |
| PPS | Per protocol set |
| PSA | Prostate specific antigen |
| PT | Preferred term |
| RBC | Red blood cell |
| RDW | Red cell distribution width |
| RP | Radical prostatectomy |
| RRT | Radical external beam radiotherapy |
| RT | Radiotherapy |
| SAE | Serious adverse event |
| SAF | Safety analysis set |
| SAP | Statistical analysis plan |
| SD | Standard deviation |

Syne qua non study no: BLS14004

Blue Earth Diagnostics study no: BED-004

SOC System organ class

TEAE Treatment emergent adverse event
TNM TNM classification of malignant tumours

WBC White blood cell

WHO World Health Organization

WHO DDE WHO Drug Dictionary Enhanced


#### 1 INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the final protocol version dated 24<sup>th</sup> March 2015 and amendments 1-4 dated 30<sup>th</sup> November 2015, 5<sup>th</sup> April 2016, 2<sup>nd</sup> March 2017 and 4<sup>th</sup> June 2018.

The SAP describes the tables, listings and figures which will be provided upon completion of the study. The SAP will be finalised before locking the database.

The table, listing and figure shells will be supplied in a separate document.

#### 2 GENERAL PRINCIPLES

The analysis and statistical reporting will be conducted at Syne qua non using SAS version 9.2 or higher.

All listings will be based on all enrolled subjects unless specified otherwise. All tables will be presented by site and overall for the appropriate analysis population.

Descriptive summary statistics for continuous variables will include number of subjects (n), mean, standard deviation (SD), minimum, median, and maximum, unless specified otherwise. The precision of these summary statistics is defined in the table, figure and listing shells document.

Descriptive summary statistics for categorical variables will include frequency counts and percentages [n (%)]. Unless stated otherwise, the denominator for percentage calculations will be the number of subjects in the analysis set.

For treatment response baseline prostate specific antigen (PSA) is the most recent PSA measurement prior to salvage therapy for subjects who had salvage treatment and the most recent PSA measurement prior to the 18F-fluciclovine positron emission tomography/computerised tomography (PET/CT) for non-salvage subjects. If no PSA measurement is available just prior to salvage therapy, baseline will be defined as the most recent PSA measurement prior to fluciclovine (<sup>18</sup>F) scan. For all other variables, and for baseline PSA other than for treatment response, baseline is defined as the most recent value prior to fluciclovine (<sup>18</sup>F) administration.

In general, there will be no imputation of missing data, however where dates are partially missing dates may be imputed for calculation purposes, details are given under relevant section.

#### 3 STUDY OBJECTIVES AND DESIGN

### 3.1 Study Objectives

The primary objective of the study is to confirm the clinical benefit of fluciclovine (<sup>18</sup>F) PET/CT in affecting management decisions in subjects with biochemical recurrence (BCR) being considered for radical salvage treatment (with curative intent).

The secondary objectives of the study are

 To assess possible improvement in outcome of radical salvage treatment based on fluciclovine (<sup>18</sup>F) PET/CT being included in the assessment


- To assess the PSA threshold for positive lesion detection by fluciclovine (<sup>18</sup>F) PET/CT in BCR
- To assess the safety of fluciclovine (<sup>18</sup>F) injection in subjects undergoing PET/CT

# 3.2 Study Design

This will be an open-labelled, multi-centred study in the United Kingdom.

The study group will include up to 180 subjects with a diagnosis of BCR of previous radically treated prostate cancer (PCa), and who are being considered for radical salvage therapy.

Subjects will have a fluciclovine (<sup>18</sup>F) PET/CT scan in addition to standard work-up for radical salvage therapy. The clinical utility of fluciclovine (<sup>18</sup>F) PET/CT will be assessed by recording changes to the recommended management plan influenced by the scan result.

The summary flow chart of the study design is as follows:



#### 3.3 Visit Structure

The visit structure and scheduled assessments are detailed in Appendix A: Schedule of study procedures of the protocol.


### 3.4 Sample Size

For the primary objective of treatment change evaluation, a minimum of 171 subjects with complete primary endpoint data will be required to allow for a width of +/-6% in a two-sided 95% confidence interval (CI). This is based on the conservative assumption that 20% of subjects will have a treatment change, as fluciclovine (<sup>18</sup>F) PET/CT has been shown to upstage 25.7% of subjects with recurrent prostate cancer, and also based on the management change studies reported on choline PET/CT. The aim is to recruit 180 subjects for this trial, based on an anticipated primary endpoint drop-out rate of 5%.

### 3.5 Changes from the Protocol Planned Analysis

The protocol specified "Improvement in outcome of radical salvage treatment based on fluciclovine (18F) PET/CT being included in the assessment" as a secondary endpoint. This was to be assessed based on PSA and radiological response. Due to lack of data being recorded for radiological response this definition was not used, treatment response was instead assessed using PSA only (see section 5.4.2.1.).

#### 4 STUDY SUBJECTS

### 4.1 Analysis sets

The list of subjects to be included in each of the analysis set is to be agreed between the Syne qua non statistician and Blue Earth Diagnostics once all study data are available and prior to database lock.

Enrolled Set: All subjects who entered screening.

**Safety Analysis Set (SAF)**: All subjects who have been included in the database and have been administered fluciclovine (<sup>18</sup>F) will be included in the Safety Analysis Set (SAF).

**Full Analysis Set (FAS)**: All subjects enrolled who have had a fluciclovine (<sup>18</sup>F) PET/CT scan will be included in the Full Analysis Set (FAS).

**Evaluable Analysis Set (EAS)**: All subjects from the FAS who have an intended treatment management plan completed and a revised management plan page completed will be included in the Evaluable Analysis Set (EAS).

**Per Protocol Set (PPS)**: All subjects in the EAS without major significant deviation following review of the protocol deviation list.

# 4.2 Disposition of Subjects

The number and percentage of all subjects enrolled, included in each analysis set, who completed the study and who prematurely withdrew, including a breakdown of the primary reasons for withdrawal, will be presented.

All enrolled subjects will be listed indicating their membership to the evaluable analysis set along with the reason for exclusion.

Completion and withdrawal information will be listed, including individual reasons for withdrawal.


#### 4.3 Protocol Deviations

Failed inclusion criteria and failed exclusion criteria will be listed for screening failures.

The number and percentage of subjects within each deviation category will be presented by deviation type (Major Significant, Major or Minor) and by site and overall. The deviation category and type will be provided by Blue Earth Diagnostics. All protocol deviations will be listed.

## 4.4 Background and Demographic Characteristics

#### 4.4.1 Demographic and Baseline Characteristics

Demographic characteristics (age, ethnic origin and race collected at Screening), body measurements (height, weight collected, and BMI derived at Visit 2) will be summarised for the enrolled set, FAS, EAS and PPS populations.

Body mass index (BMI) is calculated as (weight (kg)/height (m)<sup>2</sup>).

Individual demographic characteristics and body measurements data will be listed.

#### 4.4.2 Medical History

Medical history events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 18.1.

The number and percentage of subjects from the FAS with previous medical history and current events will be tabulated by system organ class (SOC), preferred term (PT). SOCs will be ordered in decreasing frequency of the total number of subjects with medical history events reported in each SOC and PTs will be ordered within a SOC in decreasing frequency of the total number of subjects with each medical history event. This table will be repeated for all events, regardless of whether previous or current events.

All medical history events will be listed.

#### 4.4.3 Prostate Cancer History

Details of prostate cancer history will be summarised for subjects from the FAS, and will consist of:

- Time since initial diagnosis (months), calculated as [12\*(date of informed consent date of initial prostate cancer diagnosis + 1)/365.25]
- TNM stage: Pathological TNM stage if available, otherwise Clinical TNM stage. A summary for T1 total, T2 total and T3 total will be provided as the sum of the number of subjects in each of the subgroups plus any subjects where only T1, T2 or T3 was recorded.
- Gleason total score: Gleason total score from surgery if available, otherwise Gleason total score from biopsy
- Time since adjuvant treatment (months), calculated as [12\*(date of informed consent stop date of adjuvant treatment + 1)/365.25]
- Duration of adjuvant treatment (months), calculated as [12\*(stop date of adjuvant treatment – start date of adjuvant treatment + 1)/365.25]

- Time since diagnosis of biochemical recurrence (days), calculated as (date of informed consent – date of diagnosis of biochemical recurrence + 1). Time since diagnosis of BCR may be derived in months if more appropriate.
- Baseline PSA value
- Baseline PSA category (0 0.2, >0.2 0.5, >0.5 1, >1 2, >2 5, >5 10 and >10)

In addition, summary table to summarise baseline Prostate Specific Antigen (PSA) by Prior Radical Prostatectomy status (Prior Radical Prostatectomy vs No Prior Radical Prostatectomy) using descriptive statistics (number of subjects (n), mean, standard deviation (SD), minimum, median, and maximum), will be produced.

Details of prostate cancer history will be listed.

Date imputation for incomplete dates:

- If day part missing, put 15<sup>th</sup> of the month
- If day and month parts missing, put 01 July

#### 4.4.4 Cancer Therapies for Prostate Cancer

Cancer therapies for prostate cancer will be coded according to the World Health Organization Drug Dictionary Enhanced (WHO DDE) (Enhanced) version Sep 2015.

Cancer therapies will be categorised as follows:

Subjects with radical prostatectomy:

- Radiotherapy
- No radiotherapy

Subjects without radical prostatectomy:

- Radiotherapy only
  - o EBRT only
  - Brachytherapy only
  - EBRT and brachytherapy
- Radiotherapy and other therapies
  - EBRT and other therapies
  - Brachytherapy and other therapies
- Other therapies

Prior cancer therapies for prostate cancer are defined as those for which the end date is prior to the date of injection of fluciclovine (<sup>18</sup>F).

Concomitant/post-scan cancer therapies for prostate cancer are defined as those with a start date on or after the injection date of fluciclovine (<sup>18</sup>F), or those with a start date before the injection date of fluciclovine (<sup>18</sup>F) but which continued with a stop on or after the injection date of fluciclovine (<sup>18</sup>F). Summaries for subjects with prior and post-scan radical prostatectomy will be presented separately.

Summary table to summarise time from <sup>18</sup>F-fluciclovine PET/CT to first post-<sup>18</sup>F-fluciclovine treatment in days using descriptive statistics (number of subjects (n), mean, SD, minimum, median, and maximum) will be provided.

If cancer therapy dates are incomplete and it is not clear whether the medication was concomitant, it will be assumed to be concomitant.

The number and percentage of subjects per category of prostate cancer therapy will be presented for all subjects from the SAF, separately for subjects with and without radical prostatectomy. This summary will be repeated for prior and concomitant cancer therapies.

All therapies for prostate cancer will be listed including type of therapy, reported therapy name, medication class, standardised medication name, dose, dose unit, route of administration, start date and end date or 'ongoing' flag, therapy comments.

#### 4.4.5 Prior and Concomitant Medications

Prior and concomitant medications will be coded according to the World Health Organization Drug Dictionary Enhanced (WHO DDE) (Enhanced) version Sep 2015.

Prior medications are defined as those for which the end date is prior to the date of injection of fluciclovine (18F).

Concomitant medications are defined as those with a start date on or after the injection date of fluciclovine (<sup>18</sup>F), or those with a start date before the injection date of fluciclovine (<sup>18</sup>F) but which continued with a stop date on or after the injection date of fluciclovine (<sup>18</sup>F).

If medication dates are incomplete and it is not clear whether the medication was concomitant, it will be assumed to be concomitant.

The number and percentage of subjects who took any medications will be presented by centre and overall by medication class, standardised medication names sorted alphabetically for all subjects from the SAF, separately for prior medications and concomitant medications.

All prior and concomitant medications will be listed including reported name, medication class, standardised medication name, indication, dose, dose unit, frequency, route of administration, start date and end date or 'ongoing' flag.

## 4.5 Administration of Investigational Product

The volume of undiluted fluciclovine, activity of fluciclovine and injection site reaction during and following fluciclovine administration will be summarised for subjects in the SAF.

#### 5 EFFICACY EVALUATION

All listings will be based on the FAS unless specified otherwise. The primary efficacy analysis will be based on the EAS and will be repeated on the PPS as a secondary analysis. The secondary efficacy analyses will be based on the FAS.


#### 5.1 **Primary Efficacy Variable**

The primary efficacy variable is the record of the revised management plan post fluciclovine (<sup>18</sup>F) PET/CT scan in comparison to the pre-scan intended management plan.

#### 5.2 **Secondary Efficacy Variables**

The secondary efficacy variables are:

- The proportion of subjects who have a sustained response to radical salvage therapy.
- PSA levels in relation to scan positivity will be analysed to determine the optimal PSA threshold for detecting recurrent PCa by fluciclovine (18F) PET/CT.

## **Definition of Region Levels**

Two main regions will be analysed, the prostate and prostate bed and the extraprostatic region.

The prostate and prostate bed include the following lesion locations:

- Prostate bed left
- Prostate bed right
- Peripheral zone left
- Peripheral zone right
- Central gland left
- Central gland right
- Left seminal vesicle
- Right seminal vesicle

The extra-prostatic regions include the following lesion locations

- Lymph nodes
  - Pelvic lymph nodes
    - Common iliac left
    - Common iliac right
    - Internal iliac left
    - Internal iliac right
    - External iliac left
    - External iliac right
    - Obturator left
    - Obturator right
    - Pre-sacral left

- Pre-sacral right
- Peri-rectal anterior
- Peri-rectal posterior
- Peri-rectal left
- Peri-rectal right
- Inguinal left
- Inguinal right

Date: 10OCT2018 Version: Amendment 1 Final ST/form/010/6

- Retroperitoneal lymph nodes
  - Para-aortic
  - Retro-aortic
  - Para-caval
  - Retro-caval
- Other lymph nodes
  - Intra-peritoneal
  - Mediastinal left
  - Mediastinal right
  - Axillary left
- Soft tissues/parenchyma
  - o Lung upper lobe left
  - Lung upper lobe right
  - Lung middle lobe right
  - Lung lower lobe left
  - o Lung lower lobe right
  - Brain left
  - o Brain right
  - Liver left
  - Liver right
  - Spleen
  - Subcutaneous/cutaneous
  - Muscle
  - Bowel
- Bones
  - o Skull
    - Skull base/maxilla left
    - Skull base/maxilla right
    - Mandible left
    - Mandible right
  - Vertebra
    - Vertebra C1
    - Vertebra C2
    - Vertebra C3
    - Vertebra C4

- Aorto-caval
- Retrocrural left
- Retrocrural right
- Axillary right
- Cervical left
- Cervical right

Vertebra C5

Vertebra C6

Vertebra C7

Vertebra T1

Date: 10OCT2018 Version: Amendment 1 Final ST/form/010/6

- Vertebra T2
- Vertebra T3
- Vertebra T4
- Vertebra T5
- Vertebra T6
- Vertebra T7
- Vertebra T8
- Vertebra T9
- Vertebra T10
- Vertebra T11

#### o Chest

- 1<sup>st</sup> rib left
- 1st rib right
- 2<sup>nd</sup> rib left
- 2<sup>nd</sup> rib right
- 3<sup>rd</sup> rib left
- 3<sup>rd</sup> rib right
- 4<sup>th</sup> rib left
- 4<sup>th</sup> rib right
- 5<sup>th</sup> rib left
- 5<sup>th</sup> rib right
- 6<sup>th</sup> rib left
- 6<sup>th</sup> rib right
- 7<sup>th</sup> rib left
- 7<sup>th</sup> rib right
- 8<sup>th</sup> rib left

#### Pelvis

- Ilium left
- Ilium right
- Superior pubic ramus left
- Superior pubic ramus right
- Inferior pubic ramus left

- Vertebra T12
- Vertebra L1
- Vertebra L2
- Vertebra L3
- Vertebra L4
- Vertebra L5
- Sacrum left
- Sacrum right
- Sacrum central
- 8<sup>th</sup> rib right
- 9<sup>th</sup> rib left
- 9<sup>th</sup> rib right
- 10<sup>th</sup> rib left
- 10<sup>th</sup> rib right
- 11<sup>th</sup> rib left
- 11<sup>th</sup> rib right
- 12<sup>th</sup> rib left
- 12<sup>th</sup> rib right
- Sternum
- Clavicle left
- Clavicle right
- Scapula left
- Scapula right
- Inferior pubic ramus right
- Pubic body left
- Pubic body right
- Ischium left
- Ischium right

Version: Amendment 1 Final ST/form/010/6

### Appendicular

- Proximal humerus left
- Proximal humerus right
- Proximal femur left
- Proximal femur right

## 5.4 Statistical Analysis

#### **5.4.1 Primary Efficacy Analysis**

The analysis of the primary outcome will be performed on the EAS as the primary analysis and will be repeated on the PPS as a secondary analysis. Comparisons between the original treatment plan and the revised treatment plan will be categorised as no change, major change or other change. The definitions of the change categories are listed below.

- No change: the original treatment plan is the same as the revised treatment plan
- Major change: the original treatment plan is not the same as the revised treatment plan and the grouping for the original treatment plan is not the same as the grouping for the revised treatment plan

These will be further split and presented according to the following categories:

- Salvage or Non-curative systemic therapy to Watchful waiting
- Salvage therapy to Non-curative systemic therapy
- Non-curative systemic therapy to Salvage therapy
- Alternative Major change
- Other change: the original treatment plan is not the same as the revised treatment plan but the grouping for the original treatment plan is the same as the grouping for the revised treatment plan

These will be further split and presented according to the following categories:

- Modified RT field plan
- Modified androgen-deprivation regimen
- Alternative Other change

Groupings of treatment plans are detailed in the following table:


Version: Amendment 1 Fina ST/form/010/6

| Original Treatment<br>Plan | Grouping for<br>Original Tx Plan | Revised Treatment | Grouping for<br>Revised Tx Plan |
|---|---|---|---|
| Was androgen deprivation therapy planned | Androgen<br>Deprivation<br>Therapy | Androgen deprivation therapy | Androgen<br>deprivation therapy |
| | | Watch and wait | Watch and wait |
| | | Chemotherapy | Chemotherapy |
| Salvage<br>radiotherapy to the<br>prostate bed | | Salvage radiotherapy to the prostate bed | |
| Salvage radiotherapy to the prostate bed, with boost to areas guided by conventional imaging | Salvage<br>Radiotherapy | Salvage radiotherapy to the prostate bed, with boost to areas guided by conventional imaging | Salvage<br>Radiotherapy |
| | | Salvage radiotherapy to the prostate bed with boost to areas guided by fluciclovine (18F) PET/CT | |
| Salvage<br>radiotherapy to the<br>prostate bed and<br>whole pelvis | | Salvage<br>radiotherapy to the<br>prostate bed and<br>whole pelvis | |
| Salvage radiotherapy to the prostate bed and whole pelvis, with boost to areas guided by conventional imaging | Salvage<br>Radiotherapy | Salvage radiotherapy to the prostate bed and whole pelvis, with boost to areas guided by conventional imaging | Salvage<br>Radiotherapy |
| | | Salvage radiotherapy to the prostate bed and whole pelvis with boost to areas guided by fluciclovine (18F) PET/CT | |

Date: 10OCT2018 Version: Amendment 1 Final ST/form/010/6

| Original Treatment<br>Plan | Grouping for<br>Original Tx Plan | Revised Treatment Plan | Grouping for<br>Revised Tx Plan |
|---|---|---|---|
| Salvage<br>cryotherapy | | Salvage<br>cryotherapy | |
| | Salvage<br>Cryotherapy | Salvage cryotherapy with boost to areas guided by fluciclovine (18F) PET/CT | Salvage<br>Cryotherapy |
| Salvage<br>brachytherapy | | Salvage<br>brachytherapy | |
| | Salvage<br>Brachytherapy | Salvage brachytherapy with boost to areas guided by fluciclovine (18F) PET/CT | Salvage<br>Brachytherapy |
| | | Salvage brachytherapy with treatment plan guided by fluciclovine (18F) PET/CT | |
| Salvage HIFU | | Salvage HIFU | |
| | Salvage HIFU | Salvage HIFU with treatment plan guided by fluciclovine (18F) PET/CT | Salvage HIFU |
| Salvage prostatectomy | | Salvage prostatectomy | |
| | Salvage<br>Prostatectomy | Salvage prostatectomy with targeted resection / sampling of fluciclovine (18F) positive areas outside conventional surgical field | Salvage<br>Prostatectomy |
| Salvage<br>prostatectomy and<br>limited lymph node<br>dissection | | Salvage<br>prostatectomy and<br>limited lymph node<br>dissection | |

Date: 10OCT2018 Version: Amendment 1 Final ST/form/010/6

| Original Treatment<br>Plan | Grouping for<br>Original Tx Plan | Revised Treatment<br>Plan | Grouping for<br>Revised Tx Plan |
|---|---|---|---|
| | | Salvage prostatectomy and limited lymph node dissection with targeted resection / sampling of fluciclovine (18F) positive areas outside surgical field | |
| Salvage prostatectomy and extended lymph node dissection (including internal and external iliac, and obturator nodes) | | Salvage prostatectomy and extended lymph node dissection (including internal and external iliac, and obturator nodes) | |
| | | Salvage prostatectomy and extended lymph node dissection (including internal and external iliac, and obturator nodes) with targeted resection / sampling of fluciclovine (18F) positive areas outside surgical field | |
| | | Targeted salvage treatment of fluciclovine (18F) positive extra-pelvic / bony areas | Targeted salvage<br>treatment |
| | | Other | Other |

The classification and sub-classification of change in treatment management plan will be agreed prior to data base lock.

The number, percentage and exact 95% CI of subjects with and without a change in management plan after the fluciclovine (18F) scan results become available will be presented. In addition, the number and percentage of subjects with changes categorised as major or other will be presented. These summaries will be repeated separately for subjects with a positive and a negative fluciclovine (18F) scan and for subjects without prostatectomy and with prostatectomy.

Date: 10OCT2018 Version: Amendment 1 Final ST/form/010/6

The number, percentage and 95% CI of subjects who agreed to the revised management plan after fluciclovine (<sup>18</sup>F) scan results become available will be presented.

Details of the intended management plan, revised management plan and agreed management plan will be listed.

#### 5.4.2 Secondary Efficacy Analyses

#### 5.4.2.1 Treatment response as assessed by change in PSA

An assessment of treatment response, which is based on the percentage change in PSA from baseline to the last value reported, is defined as:

- >=30% decrease in PSA will be considered to be a response to treatment
- <25% increase or <30% decrease will be classified as stable disease</li>
- >=25% increase in PSA will be classified as disease progression

See section 2 General Principles for baseline definition.

The number, percentage and exact 95% CI of subjects having a treatment response, stable disease and disease progression, as assessed by change in PSA, will be presented overall and separately for subjects in the FAS who had salvage treatment, for subjects who had non-salvage treatment, for those with a change in management plan and for subjects with no change in management plan following the <sup>18</sup>F-fluciclovine PET/CT scan. In addition, treatment response assessed by change in PSA will be summarised by disease location (local disease versus extra-prostatic disease) and treatment administered.

The percentage change in PSA from baseline to the last value reported will be summarised overall and by subjects who had a change in management plan versus those who did not have a change in management plan following the <sup>18</sup>F-fluciclovine PET/CT scan, disease location and treatment administered.

Finally, a waterfall plot of the maximum percentage reduction in PSA during the 4-8 month window will be presented on the y-axis and each subject will be represented by a bar on the x-axis. The bars will be ordered in descending order of the magnitude of the percentage change in PSA value.

Treatment response and the factors used to assess the response will be listed in full.

#### 5.4.2.2 PSA threshold

The detection rate (DR) will be calculated as number of positive fluciclovine (<sup>18</sup>F) scan results/total number of scans.


The point estimate (expressed in percentage) of the DR will be presented at the region level and at the subject level. These rates will be presented for all subjects from the FAS and PPS, overall and across a range of baseline PSA values:

- 0 0.2
- $\bullet$  >0.2 0.5
- $\bullet$  >0.5 1.0
- $\bullet$  >1.0 2.0
- $\bullet$  >2.0 5.0
- $\bullet$  >5.0 10.0
- >10.0

to determine the optimum PSA threshold for lesion detection. See section 2 General Principles for baseline definition.

The detection rates will also be summarised across the following baseline Gleason score categories: <=6, 7, 8 and >=9.

All fluciclovine (18F) and other imaging results will be listed.

#### **Handling of Dropouts or Missing Data** 5.4.3

Subjects who withdrew from the study prior to completion will be summarised. Withdrawn subjects will not be directly replaced and no imputation of missing data will be conducted.

#### 5.4.4 **Interim Analyses and Data Monitoring**

A single interim analysis of the primary endpoint will be performed in the first 85 evaluable subjects. If the number of treatment changes is greater than 45 (52.9%, with a 97.5% two-sided CI of 40.3%-62.3%, so the lower limit is over 40%), the trial will be terminated early due to overwhelming effectiveness. If the number of treatment changes is 8 or fewer (9.4%, with a 97.5% two-sided CI of 3.6%-18.9%, so the upper limit in this population is below the 20% of the null hypothesis), the trial will be terminated early due to futility.

#### **Examination of Subgroups**

No subgroup analyses will be conducted during the study.

#### **Site Specific Sub-study** 5.4.6

A site specific sub-study will be conducted in order to compare the ordered subset expectation maximisation (OSEM) standard of care method of reconstructing PET/CT images with that of the Bayesian penalised likelihood method of PET/CT image reconstruction. The analysis of the sub-study results is beyond the scope of this SAP.

#### SAFETY EVALUATION

All safety evaluations will be performed on the safety analysis set (SAF) unless specified otherwise.


All safety tables will be presented by centre and overall.

Subjects will be included and counted in summary tables only if they have available data.

### 6.1 Adverse Events

Adverse events (AE) will be coded using the Medical Dictionary for Regulatory Activities (MedDRA) version 17.1.

A treatment-emergent adverse event (TEAE) is defined as an AE with start date/time on or after the start/time of fluciclovine (<sup>18</sup>F) administration, or AEs with worsening intensity on or after the start date/time of fluciclovine (<sup>18</sup>F) administration.

AEs with unknown start date/time will be assumed to be treatment-emergent unless the end date/time is known to be before the fluciclovine (<sup>18</sup>F) administration.

Summary tables will be produced for all TEAEs occurring up to 42 days (i.e. occurring between day 1 and day 43) after the fluciclovine (<sup>18</sup>F) administration.

An overall summary of TEAEs will be created including:

- number of TEAEs and number of subjects with TEAEs,
- number of TEAEs and number of subjects with TEAEs associated with the injection site,
- number of serious TEAEs and number of subjects with serious TEAEs,
- number of subjects with TEAEs by CTCAE grade (Grade 1 to Grade 5),
- number of subjects with TEAEs by relationship to fluciclovine (unrelated, possibly related, probably related, definitely related and related, where related adverse events are those classified as possibly, probably and definitely related to fluciclovine <sup>18</sup>F)

The number and percentage of subjects experiencing TEAEs will be presented by system organ class (SOC) and preferred term (PT). System organ class and preferred term will be presented in decreasing frequency of the total number of subjects with TEAEs. If a subject experienced more than one treatment-emergent adverse event, the subject will be counted once for each system organ class and once for each preferred term.

The number and percentage of subjects experiencing TEAEs will be presented by SOC, PT and CTCAE grade. SOC and PT will be presented in decreasing frequency of the total number of subjects with TEAEs. If a subject experienced more than one TEAE, the subject will be counted once for each SOC and once for each PT at the worst severity.

The number and percentage of subjects experiencing TEAEs will be presented by SOC, PT and relationship to study drug. SOC and PT will be presented in decreasing frequency of the total number of subjects with TEAEs. If a subject experienced more than one TEAE, the subject will be counted once for each SOC and once for each PT at the closest relationship to study drug.

All adverse events will be listed and TEAEs will be identified. AEs occurring up to 42 days after fluciclovine (<sup>18</sup>F) administration will be flagged. All SAEs will be listed separately.


### 6.2 Clinical Laboratory Evaluation

### 6.2.1 Haematology

Haematology values will be summarised by parameter and visit, and also for change from baseline (last pre-scan value vs first post-scan value).

All haematology values will be listed showing reference ranges (flagging abnormal findings).

### 6.2.2 Biochemistry

Biochemistry values will be summarised by parameter and visit, and also for change from baseline (last pre-scan value vs first post-scan value).

Additionally, from the serum creatinine levels (mg/dL), creatinine clearance (CrCl) will be derived using the Cockcroft Gault formula (Cockroft DW, 1976) and the glomerular filtration rate (GFR) will be derived using the MDRD formula (Levey AS, 2006) as follows:

- Cockcroft-Gault formula: CrCl (mL/min) = [(140 age) \* (Weight in kg) \* (0.85 if female)] / (72 \* Creatinine)
- MDRD formula: GFR (mL/min) = 175 \* Creatinine<sup>-1.154</sup> \* age<sup>-0.203</sup> \* (1.212 if subject is black) \* (0.742 if female)

CrCl and GFR categories (≤30 mL/min, >30 - ≤60, >60 - ≤90, >90 mL/min) will be summarised by time window, and the shift table of baseline status against the worst status on or after fluciclovine (¹8F) administration will be presented.

All biochemistry values will be listed showing reference ranges and flagging abnormal findings.

#### 6.2.3 Urinalysis dipstick

All urinalysis results will be listed.

#### 6.2.4 Urine microscopy

All urine microscopy results will be listed.

## 6.3 Vital Signs

Vital signs include pulse rate, systolic and diastolic blood pressure.

Vital sign values will be summarised by parameter and time point, and also for change from baseline.

Details of vital signs data will be listed.

## 6.4 Electrocardiography

Electrocardiogram (ECG) interpretation is recorded at screening and visit 4.

ECG interpretations will be summarised by shift tables highlighting any changes between screening and visit 4.


#### 7 REFERENCES

- Cockroft DW, G. M. (1976). Prediction of creatinine clearance from serum creatinine. *Nephron*, 31-41.
- Levey AS, C. J. (2006). Using standardized serum creatinine values in the modification of diet in renal disease study equation for estimating glomerular filtration rate. *Ann Intern Med*, 247-254.




**Certificate Of Completion** 

Envelope Id: 93B644B8A8914520914F18451BC4D479

Subject: BED004 (BLS14004): Statistical Analysis Plan Amendment 1 for signature

Source Envelope:

Document Pages: 22Signatures: 2Envelope Originator:Certificate Pages: 5Initials: 0Elizabeth GardenerAutoNav: EnabledGostling HouseEnvelopeld Stamping: EnabledDiss Business Park

Time Zone: (UTC) Dublin, Edinburgh, Lisbon, London Diss, Norfolk IP22 4GT

elizabeth.gardener@synequanon.com

IP Address: 62.232.1.93

Sent: 10/11/2018 11:19:15 AM

Viewed: 10/11/2018 11:19:49 AM

Signed: 10/11/2018 11:20:20 AM

Sent: 10/11/2018 11:20:21 AM

Viewed: 10/11/2018 11:31:22 AM

Signed: 10/11/2018 11:31:58 AM

Status: Completed

**Record Tracking** 

Status: Original Holder: Elizabeth Gardener Location: DocuSign

10/11/2018 11:13:39 AM elizabeth.gardener@synequanon.com

Signer Events Signature Timestamp

Elizabeth Gardener

Elizabeth Gardener

elizabeth.gardener@synequanon.com

Senior Statistician Syne qua non

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

A40AC555-1C6B-49FB-A379-312B0D6DA509

Using IP Address: 62.232.1.93

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I am the author of this document

**Electronic Record and Signature Disclosure:** 

Not Offered via DocuSign

Albert Chau

albert@datacision.co.uk

Director

**Datacision Limited** 

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

albert Chan

9E0EEC5D-CDE9-44CC-ADBF-63BA0CE6CA8E

Using IP Address: 92.40.249.236

Signed using mobile

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 10/11/2018 11:31:22 AM

ID: 7c339459-f310-4678-b276-cd05df73f47d

In Person Signer Events Signature Timestamp

Editor Delivery Events Status Timestamp

Agent Delivery Events Status Timestamp

Intermediary Delivery Events Status Timestamp

| Certified Delivery Events | Status | Timestamp |
|---|---|---|
| Carbon Copy Events | Status | Timestamp |
| Corinne Hedgley Corinne.Hedgley@synequanon.com Senior Project Manager Syne qua non Ltd | COPIED | Sent: 10/11/2018 11:31:59 AM |

Security Level: Email, Account Authentication (Required)

**Electronic Record and Signature Disclosure:**Not Offered via DocuSign

| Notary Events | Signature | Timestamp |
|---|---|---|
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 10/11/2018 11:31:59 AM |
| Certified Delivered | Security Checked | 10/11/2018 11:31:59 AM |
| Signing Complete | Security Checked | 10/11/2018 11:31:59 AM |
| Completed | Security Checked | 10/11/2018 11:31:59 AM |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Syne qua non Ltd (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through your DocuSign, Inc. (DocuSign) Express user account. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to these terms and conditions, please confirm your agreement by clicking the 'I agree' button at the bottom of this document.

#### **Getting paper copies**

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. For such copies, as long as you are an authorized user of the DocuSign system you will have the ability to download and print any documents we send to you through your DocuSign user account for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. To indicate to us that you are changing your mind, you must withdraw your consent using the DocuSign 'Withdraw Consent' form on the signing page of your DocuSign account. This will indicate to us that you have withdrawn your consent to receive required notices and disclosures electronically from us and you will no longer be able to use your DocuSign Express user account to receive required notices and consents electronically from us or to sign electronically documents from us.

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through your DocuSign user account all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### **How to contact Syne qua non Ltd:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: pauline.allen@synequanon.com

#### To advise Syne qua non Ltd of your new e-mail address

To let us know of a change in your e-mail address where we should send notices and disclosures electronically to you, you must send an email message to us at Pauline.Allen@synequanon.com and in the body of such request you must state: your previous e-mail address, your new e-mail address. We do not require any other information from you to change your email address.. In addition, you must notify DocuSign, Inc to arrange for your new email address to be reflected in your DocuSign account by following the process for changing e-mail in DocuSign.

### To request paper copies from Syne qua non Ltd

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an e-mail to Pauline.Allen@synequanon.com and in the body of such request you must state your e-mail address, full name, US Postal address, and telephone number. We will bill you for any fees at that time, if any.

### To withdraw your consent with Syne qua non Ltd

To inform us that you no longer want to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your DocuSign account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may; ii. send us an e-mail to pauline.allen@synequanon.com and in the body of such request you must state your e-mail, full name, IS Postal Address, telephone number, and account number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

| Operating Systems: | Windows2000? or WindowsXP? |
|----------------------------|----------------------------------------------|
| Browsers (for SENDERS): | Internet Explorer 6.0? or above |
| Browsers (for SIGNERS): | Internet Explorer 6.0?, Mozilla FireFox 1.0, |
| | NetScape 7.2 (or above) |
| Email: | Access to a valid email account |
| Screen Resolution: | 800 x 600 minimum |
| Enabled Security Settings: | •Allow per session cookies |
| | •Users accessing the internet behind a Proxy |
| | Server must enable HTTP 1.1 settings via |
| | proxy connection |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an email message at the email address we have on file for you at that time providing you with the revised hardware and software requirements, at which time you will have the right to withdraw your consent.

#### Acknowledging your access and consent to receive materials electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please verify that you were able to read this electronic disclosure and that you also were able to print on paper or electronically save this page for your future reference and access or that you were able to e-mail this disclosure and consent to an address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format on the terms and conditions described above, please let us know by clicking the 'I agree' button below.

By checking the 'I Agree' box, I confirm that:

- I can access and read this Electronic CONSENT TO ELECTRONIC RECEIPT OF ELECTRONIC RECORD AND SIGNATURE DISCLOSURES document; and
- I can print on paper the disclosure or save or send the disclosure to a place where I can print it, for future reference and access; and
- Until or unless I notify Syne qua non Ltd as described above, I consent to receive from exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to me by Syne qua non Ltd during the course of my relationship with you.

# A Phase 3, Open-label Study to Assess the Clinical Utility of Fluciclovine (18F) PET/CT in Patients with Prostate **Cancer with Biochemical Recurrence after Radical Treatment**

Blue Earth Diagnostics Study No: BED-004 Syne qua non Ltd Study No: BLS14004

# Statistical Analysis Plan Addendum 2

**Version: Final** 

**Date: 08 March 2019** 

#### For Syne qua non Ltd - Lead Statistician

DocuSigned by: Elizabeth Gardener



Signer Name: Elizabeth Gardener

Signing Reason: I am the author of this document Signing Time: 08 March 2019 | 09:11 GMT A40AC5551C6B49FBA379312B0D6DA509

### For Blue Earth Diagnostics

DocuSigned by:

Albert Chau



Signer Name: Albert Chau Signing Reason: I approve this document Signing Time: 08 March 2019 | 09:27 GMT

9E0EEC5DCDE944CCADBF63BA0CE6CA8E

Date: 08MAR2019 Version: Addendum 2 Final

ST/form/038/1

# **Contents**

| 1 | INTRODUCTION | _ 4 |
|-----|--------------------------|-----|
| | CHANGES TO the FINAL SAP | |
| 2.1 | Change 1 | _ |
| 2.2 | Change 2 | 4 |

Date: 08MAR2019 Version: Addendum 2 Final ST/form/038/1

### **LIST OF ABBREVIATIONS**

PSA Prostate specific antigen SAP Statistical analysis plan

Date: 08MAR2019 Version: Addendum 2 Final

ST/form/038/1

#### 1 INTRODUCTION

This the second addendum to the final statistical analysis plan (SAP) Amendment 1 dated 10<sup>th</sup> October 2018, documenting additional analyses following database lock. Full details of the changes are detailed below.

### 2 CHANGES TO THE FINAL SAP

### 2.1 Change 1

Section 5.4.2.1 Treatment response as assessed by change in PSA

The number, percentage and exact 95% CI of subjects having a treatment response, stable disease and disease progression, as assessed by change in PSA, will be presented for subjects in the FAS who had salvage therapy. The summary will include an overall summary and separate summaries for subjects who had therapy guided by fluciclovine and for subjects whose therapy was not guided by fluciclovine.

This additional table will be of the same format as *Table 14.2.2.1 Treatment Response Assessment as Assessed by PSA - by Disease Location*, with the categories "Overall", "Local Disease" and "Extra-prostatic disease", replaced with "Salvage Therapy – All", "Salvage Therapy Guided by Fluciclovine" and "Salvage Therapy Not Guided by Fluciclovine" respectively.

This description is considered sufficient and a shell is not required. The title will be "Table 14.2.2.5 Treatment Response Assessment as Assessed by PSA in Subjects with Salvage Therapy - by Guided by/Not Guided by Fluciclovine".

Subjects will be determined to have a therapy guided by fluciclovine if they have an agreed therapy which contains the text string "GUIDED BY FLUCICLOVINE".

#### Reason for the change

To assess possible improvement in outcome of radical salvage treatment based on 18F fluciclovine PET/CT being included in the assessment.

## 2.2 **Change 2**

Section 5.4.2.3 Summary of disease location in subjects who had a change in management plan from salvage therapy to non-salvage therapy

The number and percentage of subjects who had positive extra-prostatic findings and negative extra-prostatic findings will be presented for subjects who had a change in management plan from salvage therapy to non-salvage therapy.

Subjects who had a change in management plan from salvage therapy to non-salvage therapy will be identified where the change of management plan is "SALVAGE THERAPY TO NON-CURATIVE SYSTEMIC THERAPY".

Positive/negative extra-prostatic findings will be determined from the imaging results.

This description is considered sufficient and a shell is not required. The title will be "Table 14.2.2.6 Presence of Extra-prostatic Disease in Subjects with Change of Management Plan from Salvage Therapy to Non-salvage Therapy".

Date: 08MAR2019 Version: Addendum 2 Final ST/form/038/1

Blue Earth Diagnostics study no: BED004

Syne qua non study no: BLS14004

### Reason for the change

This is an exploratory descriptive analysis to aid interpretation of the change in management plan data.

Date: 08MAR2019 Version: Addendum 2 Final

ST/form/038/1



**Certificate Of Completion** 

Envelope Id: 5BE13F32F6D64C38B8521A3A0545F67E

Subject: BED004 (BLS14004) Statistical Analysis Plan Amendment 2 for signature

Source Envelope:

Document Pages: 5 Signatures: 2 Envelope Originator:
Certificate Pages: 5 Initials: 0 Elizabeth Gardener
AutoNav: Enabled Gostling House
Envelopeld Stamping: Enabled Diss Business Park

Time Zone: (UTC) Dublin, Edinburgh, Lisbon, London

Diss Business Park

Diss Business Park

Diss, Norfolk IP22 4GT

elizabeth.gardener@synequanon.com

IP Address: 62.232.1.93

Sent: 08 March 2019 | 09:11

Viewed: 08 March 2019 | 09:11

Signed: 08 March 2019 | 09:11

Sent: 08 March 2019 | 09:11

Viewed: 08 March 2019 | 09:27

Signed: 08 March 2019 | 09:27

Status: Completed

**Record Tracking** 

Status: Original Holder: Elizabeth Gardener Location: DocuSign

08 March 2019 | 09:08 elizabeth.gardener@synequanon.com

Signer Events Signature Timestamp

Elizabeth Gardener

Elizabeth Gardener

elizabeth.gardener@synequanon.com

Senior Statistician Syne qua non

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

A40AC555-1C6B-49FB-A379-312B0D6DA509

Using IP Address: 62.232.1.93

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I am the author of this document

**Electronic Record and Signature Disclosure:** 

Not Offered via DocuSign

Albert Chau

albert@datacision.co.uk

Director

**Datacision Limited** 

Security Level: Email, Account Authentication

(Required)

Signature Adoption: Pre-selected Style

Signature ID:

albert Chan

9E0EEC5D-CDE9-44CC-ADBF-63BA0CE6CA8E

Using IP Address: 82.41.77.67

Signed using mobile

With Signing Authentication via DocuSign password

With Signing Reasons (on each tab):

I approve this document

**Electronic Record and Signature Disclosure:** 

Accepted: 08 March 2019 | 09:27

ID: 29a198c1-cdfb-44c3-b790-8ab73b128127

In Person Signer Events Signature Timestamp

Editor Delivery Events Status Timestamp

Agent Delivery Events Status Timestamp

Intermediary Delivery Events Status Timestamp

| Certified Delivery Events | Status | Timestamp |
|---|---|---|
| Carbon Copy Events | Status | Timestamp |
| Corinne Hedgley Corinne.Hedgley@synequanon.com Senior Project Manager Syne qua non Ltd Security Level: Email, Account Authentication (Required) | COPIED | Sent: 08 March 2019 09:27 |

**Electronic Record and Signature Disclosure:**Not Offered via DocuSign

| Notary Events | Signature | Timestamp |
|---|---|---|
| Envelope Summary Events | Status | Timestamps |
| Envelope Sent | Hashed/Encrypted | 08 March 2019 09:27 |
| Certified Delivered | Security Checked | 08 March 2019 09:27 |
| Signing Complete | Security Checked | 08 March 2019 09:27 |
| Completed | Security Checked | 08 March 2019 09:27 |
| Payment Events | Status | Timestamps |
| Electronic Record and Signature Disclosure | | |

#### ELECTRONIC RECORD AND SIGNATURE DISCLOSURE

From time to time, Syne qua non Ltd (we, us or Company) may be required by law to provide to you certain written notices or disclosures. Described below are the terms and conditions for providing to you such notices and disclosures electronically through your DocuSign, Inc. (DocuSign) Express user account. Please read the information below carefully and thoroughly, and if you can access this information electronically to your satisfaction and agree to these terms and conditions, please confirm your agreement by clicking the 'I agree' button at the bottom of this document.

#### **Getting paper copies**

At any time, you may request from us a paper copy of any record provided or made available electronically to you by us. For such copies, as long as you are an authorized user of the DocuSign system you will have the ability to download and print any documents we send to you through your DocuSign user account for a limited period of time (usually 30 days) after such documents are first sent to you. After such time, if you wish for us to send you paper copies of any such documents from our office to you, you will be charged a \$0.00 per-page fee. You may request delivery of such paper copies from us by following the procedure described below.

### Withdrawing your consent

If you decide to receive notices and disclosures from us electronically, you may at any time change your mind and tell us that thereafter you want to receive required notices and disclosures only in paper format. How you must inform us of your decision to receive future notices and disclosure in paper format and withdraw your consent to receive notices and disclosures electronically is described below.

### Consequences of changing your mind

If you elect to receive required notices and disclosures only in paper format, it will slow the speed at which we can complete certain steps in transactions with you and delivering services to you because we will need first to send the required notices or disclosures to you in paper format, and then wait until we receive back from you your acknowledgment of your receipt of such paper notices or disclosures. To indicate to us that you are changing your mind, you must withdraw your consent using the DocuSign 'Withdraw Consent' form on the signing page of your DocuSign account. This will indicate to us that you have withdrawn your consent to receive required notices and disclosures electronically from us and you will no longer be able to use your DocuSign Express user account to receive required notices and consents electronically from us or to sign electronically documents from us.

#### All notices and disclosures will be sent to you electronically

Unless you tell us otherwise in accordance with the procedures described herein, we will provide electronically to you through your DocuSign user account all required notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to you during the course of our relationship with you. To reduce the chance of you inadvertently not receiving any notice or disclosure, we prefer to provide all of the required notices and disclosures to you by the same method and to the same address that you have given us. Thus, you can receive all the disclosures and notices electronically or in paper format through the paper mail delivery system. If you do not agree with this process, please let us know as described below. Please also see the paragraph immediately above that describes the consequences of your electing not to receive delivery of the notices and disclosures electronically from us.

#### **How to contact Syne qua non Ltd:**

You may contact us to let us know of your changes as to how we may contact you electronically, to request paper copies of certain information from us, and to withdraw your prior consent to receive notices and disclosures electronically as follows:

To contact us by email send messages to: pauline.allen@synequanon.com

#### To advise Syne qua non Ltd of your new e-mail address

To let us know of a change in your e-mail address where we should send notices and disclosures electronically to you, you must send an email message to us at Pauline.Allen@synequanon.com and in the body of such request you must state: your previous e-mail address, your new e-mail address. We do not require any other information from you to change your email address.. In addition, you must notify DocuSign, Inc to arrange for your new email address to be reflected in your DocuSign account by following the process for changing e-mail in DocuSign.

### To request paper copies from Syne qua non Ltd

To request delivery from us of paper copies of the notices and disclosures previously provided by us to you electronically, you must send us an e-mail to Pauline.Allen@synequanon.com and in the body of such request you must state your e-mail address, full name, US Postal address, and telephone number. We will bill you for any fees at that time, if any.

### To withdraw your consent with Syne qua non Ltd

To inform us that you no longer want to receive future notices and disclosures in electronic format you may:

i. decline to sign a document from within your DocuSign account, and on the subsequent page, select the check-box indicating you wish to withdraw your consent, or you may; ii. send us an e-mail to pauline.allen@synequanon.com and in the body of such request you must state your e-mail, full name, IS Postal Address, telephone number, and account number. We do not need any other information from you to withdraw consent.. The consequences of your withdrawing consent for online documents will be that transactions may take a longer time to process..

#### Required hardware and software

| Operating Systems: | Windows2000? or WindowsXP? |
|----------------------------|----------------------------------------------|
| Browsers (for SENDERS): | Internet Explorer 6.0? or above |
| Browsers (for SIGNERS): | Internet Explorer 6.0?, Mozilla FireFox 1.0, |
| | NetScape 7.2 (or above) |
| Email: | Access to a valid email account |
| Screen Resolution: | 800 x 600 minimum |
| Enabled Security Settings: | •Allow per session cookies |
| | •Users accessing the internet behind a Proxy |
| | Server must enable HTTP 1.1 settings via |
| | proxy connection |

<sup>\*\*</sup> These minimum requirements are subject to change. If these requirements change, we will provide you with an email message at the email address we have on file for you at that time providing you with the revised hardware and software requirements, at which time you will have the right to withdraw your consent.

#### Acknowledging your access and consent to receive materials electronically

To confirm to us that you can access this information electronically, which will be similar to other electronic notices and disclosures that we will provide to you, please verify that you were able to read this electronic disclosure and that you also were able to print on paper or electronically save this page for your future reference and access or that you were able to e-mail this disclosure and consent to an address where you will be able to print on paper or save it for your future reference and access. Further, if you consent to receiving notices and disclosures exclusively in electronic format on the terms and conditions described above, please let us know by clicking the 'I agree' button below.

By checking the 'I Agree' box, I confirm that:

- I can access and read this Electronic CONSENT TO ELECTRONIC RECEIPT OF ELECTRONIC RECORD AND SIGNATURE DISCLOSURES document; and
- I can print on paper the disclosure or save or send the disclosure to a place where I can print it, for future reference and access; and
- Until or unless I notify Syne qua non Ltd as described above, I consent to receive from exclusively through electronic means all notices, disclosures, authorizations, acknowledgements, and other documents that are required to be provided or made available to me by Syne qua non Ltd during the course of my relationship with you.